CLINICAL TRIAL: NCT03044418
Title: Anesthesia of Endolaryngeal Surgery With a Special Endotracheal Laser Tube
Brief Title: Anesthesia With Endotracheal Laser Tube
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Timea Bocskai, Principal Investigator, University of Pecs
Other Study IDs: 6419
Record Dates: First submitted 2017-01-29; First posted 2017-02-07 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; Anesthesia Morbidity
Keywords: laser; endotracheal tube; total intravenous anesthesia; side effect; endolaryngeal surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesia with laser tube: The special endotracheal (ET) laser tube is tested during endolaryngeal laser surgery. Anesthesia type is the total intravenous anesthesia with propofol. We tested the application of ET laser tube in propofol anesthesia.
  Interventions: Other: Application of ET laser tube in propofol anesthesia

INTERVENTIONS:
Other: Application of ET laser tube in propofol anesthesia — The special ET laser tube covered by aluminum tape is used during anesthesia of endolaryngeal laser surgery.

SUMMARY:
The study examines the special endotracheal laser tube during anesthesia of endolaryngeal laser surgery.

DETAILED DESCRIPTION:
The special endotracheal tube is covered by a special aluminum tape.

ELIGIBILITY:
Inclusion Criteria:

* laser surgery

Exclusion Criteria:

* allergy of propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with endolaryngeal laser surgery and after 18 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Bogar, MedHabil, Study Chair — PTE Department of the Anesthesiology and Intensive Therapy; Laszlo Lujber, PhD, Study Chair — PTE Department of ENT
Locations (1):
- PTE Department of ENT, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Anesthesia With Special ET Laser Tube: The special ET laser tube is tested during endolaryngeal laser surgery. Anesthesia type is the total intravenous anesthesia with propofol. We test the application of ET laser tube in propofol anesthesia.
  The special endotracheal laser tube covered by aluminum tape is used during anesthesia of endolaryngeal laser surgery.
Period: Overall Study
Arm/Group | Anesthesia With Special ET Laser Tube
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- The Side Effects of Anesthesia With Special ET Laser Tube: The frequency of side effects of anesthesia with a special ET laser tube is tested during endolaryngeal laser surgery. Anesthesia type is the total intravenous anesthesia with propofol. We test the application of ET laser tube in propofol anesthesia.
  The special endotracheal laser tube covered by aluminum tape is used during anesthesia of endolaryngeal laser surgery.
Arm/Group | The Side Effects of Anesthesia With Special ET Laser Tube
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants] — adults over 18 years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 30
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants] — Etnicity of patients was European.
  participants
    European | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Effects
Description: problem with airway or special laser tube
Time Frame: 5 months
Measure: Number; unit: participants
Groups:
- Anesthesia With Laser Tube: the side effects of anesthesia with a special ET laser tube
Arm/Group | Anesthesia With Laser Tube
Number analyzed (Participants) | 30
participants | 0

ADVERSE EVENTS:
Time Frame: 6 months; between January 2017 and June 2017 during our study
Groups:
- The Frequency of Side Effects of Special ET Laser Tube Using: The frequency of side effects of anesthesia with special ET laser tube are analysed during endolaryngeal laser surgery. Anesthesia type is the total intravenous anesthesia with propofol. We tested the application of ET laser tube in propofol anesthesia.
  The special endotracheal laser tube covered by aluminum tape is used during anesthesia of endolaryngeal laser surgery.
Arm/Group | The Frequency of Side Effects of Special ET Laser Tube Using
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
The special laser tube is used only for less than one hour

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03044418/Prot_000.pdf